CLINICAL TRIAL: NCT06845969
Title: Reducing Dangerous Placement of Needles by Physiotherapists Who Use Dry Needling (DN) by Introducing Cadaver Anatomy Review: a Randomized Control Trial Assessing Needle Placement Accuracy and Confidence
Brief Title: Physiotherapy Dry Needling Accuracy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00128708
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Dry Needling; Physiotherapy
Keywords: Dry Needling; Safety; Accuracy; Physiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education: dry needling theory (Sham Comparator): A two hour on-line synchronous educational model focused on dry needling theory.
  Interventions: Other: Education: dry needling theory
- Education: Cadaver anatomy review (Experimental): A two hour cadaver lab review course focused on high risk areas for dry needling.
  Interventions: Other: Education: Cadaver anatomy review

INTERVENTIONS:
Other: Education: dry needling theory — Education relating to the theory of dry needling by physiotherapists
  Arms: Education: dry needling theory
Other: Education: Cadaver anatomy review — Educational instruction regarding the safe implementation of dry needling by physiotherapists using cadaver material.
  Arms: Education: Cadaver anatomy review

SUMMARY:
The goal of this clinical trial is to learn if the addition of cadaver review improves:

* the accuracy of physiotherapists who practice dry needling.
* the perceived safety of dry needling by physiotherapists. Researchers will compare the effects of an anatomy review using cadaver material to that of an educational intervention not related to anatomy to see if the anatomy review improves the needling accuracy and safety of physiotherapist who practice dry needling as compared to the control intervention of education not related to anatomy.

Participants will:

* Needle three muscles related to safety and/or accuracy using ultrasound imaging to gather accuracy and safety measurements.
* Take an initial knowledge exam capturing their knowledge on needling safety.
* Be randomized into a control group or intervention group.
* The control group will receive an online educational session not related to anatomy.
* The intervention group will receive a cadaver anatomy review class focused on high-risk area.
* Re-take a knowledge exam after their course (either cadaver lab or on-line education) to capture any change.
* Needle the same three muscles again using ultrasound to capture accuracy and safety measurements.

If reviewing anatomy using cadaver materials improve physiotherapists needling accuracy and safety, then this educational intervention could be recommended to be added to dry needling course instruction.

DETAILED DESCRIPTION:
Objectives: To determine if offering additional cadaver anatomy training focusing on high-risk areas improves needle placement accuracy and affects confidence of physiotherapists who practice dry needling compared to education focused on DN techniques.

Methods Study design: Parallel Randomized Controlled Trial (following CONSORT reporting guidelines)

Sample:

Physiotherapists: Sixty physiotherapists will be recruited consecutively using advertising in the College and Association newsletters, social media and through private physiotherapy clinics.

Needled participants: Advertisement for needled participants will be done using the same strategies above as well as through the acupuncture program at Grant MacEwan University. This will help ensure that the needled participants recruited have experience with receiving needling treatments prior to the study.

To control for variability in needling participants between therapists as well as between groups, needled participants will be randomly assigned to therapists. In addition, all attempts will be made to present both a male and female needled participant for each therapist both pre and post intervention.

Procedure overview: First DN participants will complete a survey to collect baseline data and an initial online exam to capture their current level of anatomical knowledge. Initial DN accuracy measurements will be taken three separate times on three separate muscles on both sides of the body on two separate needling volunteers (ideally a male and female) using ultrasound imaging. Self-confidence in needling ability will be captured using a visual analogue scale. Then participants will be randomized to either the intervention or the control group. The intervention group will receive an interactive cadaver review class focused on high-risk areas whereas the control group will receive an online education session of the same duration based on DN techniques but devoid of anatomy instruction. Both groups will be re-tested on their anatomy by completing an on-line knowledge exam similar to the first but different enough to avoid recall. Within two weeks of completing their intervention, both groups will be re-tested for DN accuracy on the same muscles in the same manner as before and a second self-confidence estimation will be gathered using a visual analogue sale.

Baseline assessment:

Needling Physiotherapists: A baseline survey of the enrolled therapists will capture the following: 1. sex, 2. gender, 3. physiotherapy degree(s) and program where obtained, 4. if cadaver training was offered in their program, 5. DN granting program, 6. years of full-time experience in physiotherapy practice, 7. years of full-time experience of DN practice, 8. practice setting and 9. estimates of percentage of time of DN use and estimate the percentage that the physiotherapists needled the identified muscles used in this study in the last year (upper fibers trapezius, rhomboids and supinator). Although there are many areas of high-risk, these were chosen as these regions are most commonly associated with injury or challenge accuracy. Other areas such as suboccipitals, scalenes and sternocleidomastoid, while still considered high risk, are not universally taught, and therefore not selected in this study. At baseline and within 24 hours after receiving the allocated education programs, participants will also complete an exam to capture their current level of anatomy knowledge. This exam will include aspects of the control group educational content along with some basic DN questions to help prevent participants from understanding the scope of both interventions. Survey and exam results will be piloted with research colleagues and experienced dry needlers and administered online using REDCAP.

Pre and post training assessments Ultrasound evaluation of DN accuracy: At baseline and within 2 weeks post-intervention, therapists will be asked to insert a solid filament needle three times into the upper fibers of trapezius, rhomboids and supinator on one side on two separate needled participants. Using two separate needled participants will ensure that bilateral needling accuracy can be assessed while avoiding concerns raised in the literature about bilateral pneumothorax injuries. Therapist will be allowed to use the technique taught during the DN certification completed, which will also be recorded.

The examiner will either be a trained sonographer or be trained by a radiologist to use a B-mode curvilinear ultrasound transducer to visualize the shortest distance between any part of the needles and midpoint of the target muscle as well as the tissues at risk. A frequency of 2-5Hz will be used as this is suggested for imaging of the tissue depth of the muscles of interest and the transducer will be held perpendicular to the needle shaft so as to visualize the entire needle as recommended by Malanga and Mautner in 2014. Warm sterile gel will be used as clean needling techniques will be enforced. Sterile technique is not needed as needling into joint spaces or bursa will not occur and the participants are not immunocompromised. The Ultrasound examiner will be blinded to the education group each therapist is assigned to. Therapists inserting the needles will be blinded to the ultrasound imaging obtained during these insertions.

Ultrasound imaging has been successfully used to identify needle placement in areas of high risk and has very high intra-evaluator reliability (ICC 0.98-0.99) and good to high inter-evaluator reliability (ICC 0.79-0.93) for the thickness of muscle tissue. For example, measurements of skin to rib distance using Ultrasound measurements have been found to have adequate intertester reliability with an ICC ranging from 0.92 to 0.98 and a standard error of measurement not exceeding 10% of the maximum possible depth. Ultrasound is a safe, non-ionizing imaging technology that can be used repeatedly with metal implants, is cost effective, portable, clinically accessible and has real-time scanning capabilities. Ultrasound imaging of muscles has been validated through comparisons to MRIs (cross sectional area, muscle length and width with regression coefficients of 0.808 to 1.054), demonstrating that measurements were very satisfactory

. Self-report of confidence in placing the needle: As both accuracy and safety wil be monitored in this study, the therapist will be asked to report the level of confidence that the needles inserted remained a safe distance of less than 80% of the dangerous depth and the level of confidence that the target tissue was reached (mid-belly of the selected muscle). A study by Cushman et al. 2021, demonstrated that therapist self-reported confidence levels of safe needling using the rib as a bony backdrop did not correlate to accuracy (p = 0.153) with 24% of confident palpations being inaccurate. Therapists' self-confidence levels will be recorded using a 10- point visual analogue scale (VAS) from 0 (no confidence) to 10 (completely confident).

Post intervention: Within 24 hours after intervention, a second exam will be administered to capture any change in anatomy knowledge. This exam will cover the same content as the pre-intervention exam, but be different enough to avoid recall bias. This second exam will be compared to the baseline exam to determine gains in anatomy knowledge post intervention and to help interpret whether variability in needling accuracy is related to this new anatomy knowledge. Self confidence in needling accuracy and safety will also be recaptured using a VAS. Needle placement accuracy will be retested using the above noted ultrasound imaging within 2 weeks after participants complete their education intervention. The same number of subjects and the same muscles will be used in the reassessment of accuracy but subjects will be different from first needling assessment and the order of muscles needled will be randomized.

Needled Subject Safety: The needling procedures being imaged are not outside the scope of practice for physiotherapist who are qualified to DN and are done regularly in a clinical setting. However, as the needling procedures used in this study are considered higher-risk areas, the following precautions have been taken to ensure subject safety; 1. Due to concerns of bilateral pneumothorax in the literature, two needled participants will be provided for thoracic needling to ensure no single participant is needled bilaterally on the thorax, 2. An emergency action plan will be developed to mitigate any adverse events such as bleeding, syncope and pneumothorax, 3. To ensure no major adverse events such as pneumothorax occur, the US examiner will be instructed to stop the therapist from progressing the needle when the needle tip reaches 80% of the dangerous depth to the high-risk structure. While sharing when needle tips reach dangerous distances corresponds to giving feedback on accuracy, sharing when dangerous distance happen prioritizes ensuring safety of needled participants. Sharing when dangerous distances are observed will still allow comparing the measured accuracy as the needling depth in those instances will be recorded as 80% of the dangerous depth.

Stratification and Randomization:

Randomization: After baseline measurements, therapists will be randomized 1:1 to the intervention or the control group. Randomization will be performed electronically by the coordinator using REDCAP to maintain concealed allocation and will be stratified based on, DN experience (within 5 years of graduation vs. 5 or more, DN certification and sex). Randomly ordered block sizes of 2, 4, 6 will be used to maintain balanced groups throughout while preventing team members or patients to guess where the next participant will be allocated.

Interventions:

Experimental group: The cadaver anatomy education interventions will be informed by engaging therapists-partners, DN educators and by conducting a literature review. Among other high-risk areas, the following areas will be reviewed as they pertain directly to the outcomes of our study; upper fiber trapezius, and rhomboids have been implicated more commonly in adverse events and supinator, although not a muscle often reported in adverse events, may represent a challenge for accuracy. Therapists assigned to the intervention group will participate in group cadaver anatomy review of high-risk areas in the anatomy lab by a qualified anatomy instructor. Based on consultation with content experts (Dr. Livy and Nadine Crocker) a 2-hour cadaver review demonstrating relevant muscles in relation to high-risk areas including interactive participation, exercises and discussion in the anatomy lab is planned. The size of the group will reflect the average size of a dry needling class (n=15), additionally personal experience has demonstrated that more than 20 students per instructor in the cadaver lab becomes somewhat problematic as there is limited space around specimens for viewing and instruction.

Sham comparator group: Therapists assigned to the control group will be comparable in size and receive the same number of hours of training but delivered as online interactive educational session by the same instructor on the various types/theories of DN reviewing the advantages and disadvantages of each. Content for this intervention will be informed by a review of the literature as well as with consultation from course providers. This training controls for the possible effect of receiving any training related to the approach and attention from an expert instructor.

Methods to avoid pitfalls: To control for bias, the following strategies are implemented: 1) Randomization will be stratified for the number of DN years of experience, course provider and sex. 2) Randomization should ensure balance of known and unknown confounders between groups. 3) Evaluator will be blinded to the allocated groups. 4) Therapists will not know which subjects will be selected for needle insertions and will be tested on both a male and female subject in randomized order. 5) The instructor will not be involved in assessments. 6) The researcher reviewing ultrasound imaging for accuracy will be blinded to group allocation. 7) By using a control education program, participants are also blinded to the purpose of the study, and the study controls for the attention bias by giving the same amount of attention by the same instructor. 8) This study will attempt to recruit some of the therapists who participate in this study to be needled participants in case of low enrollment of needled participants as physiotherapists trained to dry needled are familiar with the practice and with the effects of DN.

Statistics:

Descriptive statistics will be used to describe the training and experience of the therapists. Needling accuracy measurements at baseline and after training will be compared between groups using a group by time mixed-effect model ANOVA for each at-risk site assessed. Similarly, confidence ratings for each site will be compared using the same type of mixed-effect ANOVA models. Bonferroni post-hoc tests will be performed to detect significant pairwise comparisons. Support from the University of Alberta Rehabilitation Research Center statistical consultant is available for this PhD project.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapy volunteers: Physiotherapists who are in good standing with their regulatory College and licensed to practice dry needling.
* Needling volunteers (those who will be needled) must be able to provide informed consent

Exclusion Criteria:

* Physiotherapy volunteers: Physiotherapists who are not in good standing with their regulatory College or not licensed to practice dry needling or have taken a cadaver review class post-graduation from their entry to practice physiotherapy program.
* Needling volunteers (those who will be needled): Anyone who posses any contraindications to dry needling or not within normal BMI measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Dry needling accuracy | This measurement will be taken initially when the subject enrolls in the study (Baseline) and again within two weeks of having received the intervention (either control or experimental) (Follow-up).
  The distance in millimeters between the end of the needle tip when the physiotherapist states that they believe that the needle is positioned mid-belly of the target tissue measured to the actual mid belly location of the target tissue.

SECONDARY OUTCOMES:
Dry needling safety | This measurement will be taken initially when the subject enrolls in the study (Baseline) and again within two weeks of having received the intervention (either control or experimental) (Follow-up).
  A measurement in millimeters will be taken between the end of the needle tip when the physiotherapist has stated that they believe that the needle is positioned mid belly of the target muscle to any structure at risk (lungs, organs). The shortest distance to a structure at risk is recorded.
Self-reported Confidence in needle placement | This measurement will be taken initially when the subject enrolls in the study (Baseline) and again within two weeks of having received the intervention (either control or experimental) (Follow-up).
  A self-reported perceived confidence that the needle was placed to mid-belly of the targetted muscle using a visual analague scale from 0 to 10 where 10 indicates best possible confidence.
Knowledge exam score (anatomy) | This measurement will be taken initially when the subject enrolls in the study (Baseline) and again within two weeks of having received the intervention (either control or experimental) (Follow-up).
  Total score reported out of 100% related to the anatomy knowledge assessed using the parallel forms knowledge exams assessing the anatomy knowledge and the knowledge related to dry needling theory.
Knowledge exam score (Dry Needling) | This measurement will be taken initially when the subject enrolls in the study (Baseline) and again within two weeks of having received the intervention (either control or experimental) (Follow-up).
  Total score reported out of 100% related to the dry needling knowledge assessed using the parallel forms knowledge exams assessing the anatomy knowledge and the knowledge related to dry needling theory.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Parent, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be shared either as supplement when publishing the results or deposited in the ERA (online thesis repository at University of Alberta) with the PHD thesis completed during this project.